CLINICAL TRIAL: NCT02745301
Title: Urinary Biomarkers in the Detection of Urothelial Carcinoma of the Bladder
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Element Diagnostics (Unknown)
Responsible Party: Principal Investigator, Kristen Scarpato, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 151565
Record Dates: First submitted 2015-09-18; First posted 2016-04-20 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Bladder Cancer, Biomarkers
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patient urine specimens and bladder tumor specimens
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Collection of urine and bladder tumor specimens — Voided urine (pre- and post surgical) and intraoperative bladder tumor specimens to be processed for the presence of specific biomarkers.

SUMMARY:
To assess the persistence of bladder cancer-specific biomarkers in urine collected pre-operatively, in resected cancer tissue, and in urine collected post-operatively. A panel of sensitive and specific bladder cancer biomarkers will be used to establish a signature of disease in pre-operative patients with a positive diagnosis for bladder cancer by current standard of care (e.g., in-office cystoscopy, OR cystoscopy). The specificity of these markers will be assessed, as well as the degree of non-specific signal attributable to other sources of biomolecules, by analyzing resected tumor tissue for the same biomarkers. Finally, post-operative urine will be assessed for the presence of these markers. To the extent this biomarker panel can be determined to be specific and sensitive, it may serve as an indicator of the degree to which the surgical intervention successfully eradicated the underlying disease. The investigators also aim to assess the stability of a biomarker signature in urine but evaluating several patient specimens over various time points throughout the day.

DETAILED DESCRIPTION:
Current standard of care in non-muscle invasive bladder cancer (NMIBC) relies on pathologic confirmation of negative margins as well as repeat transurethral resection. National Comprehensive Cancer Network (NCCN) and American Urological Association (AUA) guidelines specify a regular schedule of continued examination by cystoscopy and cytology to monitor the patient for the recurrence of disease.

Physicians Choice Laboratory Services (PCLS) is validating a panel of biomarkers isolated from voided urine for their combined ability to reliably detect the presence of transformed cell populations. These markers include somatic mutations in a number of oncogenes that have been well established as important etiologic factors in the development of bladder cancer in the scientific and clinical literature. In addition, regional hypermethylation of the genome is evaluated, as is the presence or absence of specific proteins involved in the disease state. Through measurement of these biomarkers using next generation sequencing and immunoassays, PCLS has been able to establish both the analytical and clinical validity of these markers in diagnosing disease. The statistical correlation of these biomarkers with the presence of transitional cell carcinoma has resulted in the ability to define a distinct disease signature indicative of disease in preliminary studies. The current study aims to expand upon these findings in an effort to offer physicians an additional tool with which to manage bladder cancer.

Hypothesis: Bladder cancer biomarkers will be elevated in preoperative and intraoperative urine specimens with direct correlation to the intact lesion(s), but will diminish significantly or disappear in urine specimens post-operatively with as a function of completion of resection. Further, the persistence of disease-specific biomarkers in urine post-operatively may correlate with the risk of recurrence or progression.

Biomarker levels will be determined from pre-, intra- and post-operative urine specimens, as well as from resected bladder tissue and will be statistically compared for changes that correlate with presence or absence of visible disease. Biomarkers from tissue samples will be quantified and compared with urine sample values.

The specific aims of the current proposal are to:

SA1): Assess the stability of a biomarker signature in urine. To date, efforts across the biomarker field have relied on the detection of cancer in the context of a single patient specimen collected at a single point in time. The consistency of the biomarker signature across specimens provided by the same patient has not been fully described. The current study will assess the consistency with which the biomarkers composing the panel can be detected across urine specimens collected at multiple points in time in a subset of patients. This data will inform the utility of single point-in-time collection with regard to accurately defining the disease signature.

SA2): Assess the persistence of bladder cancer-specific biomarkers in urine collected pre-operatively, in resected cancer tissue, and in urine collected post-operatively. A panel of sensitive and specific bladder cancer biomarkers will be used to establish a signature of disease in pre-operative patients with a positive diagnosis for bladder cancer by current standard of care (e.g., in-office cystoscopy). The specificity of these markers will be assessed, as well as the degree of non-specific signal attributable to other sources of biomolecules, by analyzing resected tumor tissue for the same biomarkers. Finally, post-operative urine will be assessed for the presence of these markers. To the extent this biomarker panel can be determined to be specific and sensitive, it may serve as an indicator of the degree to which the surgical intervention successfully eradicated the underlying disease.

SA3): Determine whether persistence of biomarkers in patient urine post-operatively correlates with recurrence or progression. The same panel of markers detected in the pre-operative urine and tumor will be assayed in voided urine collected during routine follow-up surveillance visits for a period of one year. Biomarkers will be monitored for persistence and quantitative change in levels.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed urothelial type bladder cancer
* Scheduled for a transurethral resection of bladder tumor (TURBT) or cystectomy

Exclusion Criteria:

* Less than 18 years of age
* Known concurrent upper urinary tract disease
* History of bladder or prostate radiation
* Patients who are unwilling or unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The current protocol consents and enrolls 50 patients with a diagnosis of primary or recurrent bladder cancer by cystoscopy that requires transurethral resection of the bladder tumor (TURBT) or radical cystectomy (RC). Patients will be identified for participation if known to have bladder cancer and have recurrent tumor on office cystoscopy, or may present for a new hematuria work up and have evidence of transitional cell carcinoma (TCC) on office cystoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-04; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in urinary biomarker value from baseline following removal of bladder tumor | An average of 1 month after surgery
  Urinary biomarkers will be assessed pre-operatively from voided specimens. One month post-operatively, voided urine will again be assessed for changes in the level of urinary biomarker. DNA will be isolated from tissue or urine using commercially available validated kits. DNA will be quantified by standard procedures and analyzed for somatic mutation by targeted resequencing of selected regions of the genome. Specific gene targets include TP53, FGFR3, CDKN2A, TERT, and PIK3CA. Hypermethylation analysis will be conducted by bisulfite conversion of isolated DNA and sequencing to determine degree of methylation of specific CpG islands. CpG islands located in the promoter regions of OTX1, TWIST1 and ONECUT2 will be analyzed.
  Levels of Cystatin B will be assessed by quantitative immunoassay directly from urine.

SECONDARY OUTCOMES:
Change in urinary biomarker value throughout the day | One day
  5 patients will provide and additional 2 pre-operative urine specimens (for a total of 3 preoperative specimens) from a single day to assess for any potential time-dependent variation. Each specimen must be collected at least 4 hours apart. These 5 patients will be asked to collect a "morning", "midday" and "evening" urine specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen R Scarpato, MD, Principal Investigator — Vanderbilt University
Locations (1):
- The Vanderbilt Clinic, VUMC, Nashville, Tennessee, United States

REFERENCES:
- [Background] Sjodahl G, Lauss M, Lovgren K, Chebil G, Gudjonsson S, Veerla S, Patschan O, Aine M, Ferno M, Ringner M, Mansson W, Liedberg F, Lindgren D, Hoglund M. A molecular taxonomy for urothelial carcinoma. Clin Cancer Res. 2012 Jun 15;18(12):3377-86. doi: 10.1158/1078-0432.CCR-12-0077-T. Epub 2012 May 2. PMID 22553347
- [Background] Sylvester RJ, van der Meijden AP, Oosterlinck W, Witjes JA, Bouffioux C, Denis L, Newling DW, Kurth K. Predicting recurrence and progression in individual patients with stage Ta T1 bladder cancer using EORTC risk tables: a combined analysis of 2596 patients from seven EORTC trials. Eur Urol. 2006 Mar;49(3):466-5; discussion 475-7. doi: 10.1016/j.eururo.2005.12.031. Epub 2006 Jan 17. PMID 16442208
- [Background] Cancer Genome Atlas Research Network. Comprehensive molecular characterization of urothelial bladder carcinoma. Nature. 2014 Mar 20;507(7492):315-22. doi: 10.1038/nature12965. Epub 2014 Jan 29. PMID 24476821